CLINICAL TRIAL: NCT06294652
Title: AGMT Austrian Lymphoma Registry
Status: Recruiting | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_Lymphoma_Reg
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; Diffuse large B-cel lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The Lymphoma registry will be accompanied by an optional biobanking program. Sample collection will be limited to patients that have signed an additional biobanking IC.
  The samples are taken as part of the clinical routine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Lymphomas are a group of cancers that originate in the lymphatic system, a key component of the immune system. They can be broadly categorized into two main types: Hodgkin lymphoma (HL) and non-Hodgkin lymphoma (NHL).

There are different subtypes of HL, including classical Hodgkin lymphoma (cHL) and nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL). The subtypes of cHL include nodular sclerosis, mixed cellularity, lymphocyte-rich, and lymphocyte-depleted.

Non-Hodgkin lymphomas are more diverse and comprise a wide range of subtypes, each with distinct genetic, molecular, and clinical features. Common subtypes of NHL include Diffuse large B-cell lymphoma (DLBCL), Follicular lymphoma (FL), Mantle cell lymphoma (MCL), Chronic lymphocytic leukemia (CLL), myeloma, and other rarer subgroups.

Many of these diseases typically present with lymph node enlargement, bone marrow infiltration, general and lymphoma subtype specific symptoms and laboratory abnormalities.

Novel agents have improved the prognosis of high-risk lymphoma patients in the front-line and relapsed setting and more accurate prognostic tools enable less intensive treatment for low-risk patients, while maintaining their good prognosis.

Lymphoma disease have not been systematically assessed in Austria to date. This medical registry of the AGMT is thus the first Austrian-wide standardized documentation of epidemiology, clinical course and molecular and other biologic data of this disease. As lymphomas are a very heterogeneous group, not all subtypes will always be documented simultaneously in this registry. Which lymphoma subtype is to be documented can change over time, depending on which clinical question is currently in focus.

DETAILED DESCRIPTION:
This registry is designed as international multicenter observational cohort of patients with lymphoma. Information on patient´s clinical presentation, tests, diagnosis, and treatment will be obtained through extraction of data from existing patient medical charts. Longitudinal follow-up data, including survival and tumor progression, will also be extracted from patient medical charts. This patient follow-up data will be obtained until patient death or loss to follow-up.

For documentation in the registry, no further diagnostic or therapeutic measures are required than those already necessary in general. Participation in the registry must not interfere with treatment routines. Only routine data, which has already been recorded in the patient's medical chart, is transferred to the electronic Case Report Forms (eCRF). To maintain patient confidentiality, each patient will be assigned a unique patient identifying number upon enrollment; this number will accompany the patient's medical and other registry information throughout the lifetime of the registry.

A written consent must be obtained prior to the input of data. No informed consent is required from deceased patients.

ELIGIBILITY:
Inclusion Criteria:

* The registry will include patients ≥ 18 years with lymphoma.

Exclusion Criteria:

* There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interested sites that treat patients in this indication will be invited to participate in this registry.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
General Characteristics | 10 years
  To describe general characteristics of lymphoma patients
Genetic Profiling | 10 years
  To describe genetic risk profiles
Proportion of lymphoma patients in Austria that require treatment | 10 years
  To describe the proportion of lymphoma patients in Austria that require treatment
Proportion of lymphoma patients in Austria under active surveillance | 10 years
  To describe the proportion of lymphoma patients in Austria under active surveillance
Number of patients with concomitant diseases | 10 years
  To describe concomitant diseases at diagnosis of lymphoma
Number of treatment and outcome of treatment | 10 years
  To describe treatment and outcome of treatment, among them
  * historical standard with immunochemotherapy
  * cellular therapies (e.g. Car-T cells)
  * novel immunotherapies such as bispecific antibodies
  * continuous treatment or an induction/maintenance approach
  * sequence of use of various treatments
  * treatment duration
  * treatment adjustments
  * frequency and degree of response
Patient Outcome | 10 years
  To describe patient's outcome
Toxicities | 10 years
  To describe toxicity with a focus on immunological mediated side effects of treatment (e.g. Cytokine release syndrome (CRS), Immune effector cell-associated neurotoxicity syndrome (ICAN) etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — Department of Internal Medicine III, Paracelsus Medical University Salzburg, Salzburg, Austria
Locations (1):
- Universitätsklinik für Innere Medizin III, PMU Salzburg, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No